CLINICAL TRIAL: NCT06306001
Title: Intravenous Methylene Blue for Treating Fluid-refractory, Catecholamine-resistant, Neonatal Septic Shock: a Randomized, Placebo-controlled, Superiority Trial
Brief Title: Intravenous Methylene Blue for Treating Refractory Neonatal Septic Shock
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sourabh Dutta, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIRP-2023-1820/F1
Record Dates: First submitted 2024-02-20; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Sepsis; Shock, Septic
Keywords: Methylene blue; Neonate; Septic shock; Clinical trial
MeSH Terms: conditions — Neonatal Sepsis; Shock, Septic | interventions — Methylene Blue; Saline Solution

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated to an intervention arm and a placebo arm. The 2 arms of the trial will run concurrently.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The random allocation will be concealed using serially numbered opaque sealed envelopes. After opening the envelope, a research nurse will administer a bolus of the study drug or placebo behind a screen, shielded from other staff. The infusion will be drawn up in an opaque syringe by the research nurse and infused through an intravenous tubing covered completely with aluminum foil. The research nurses will not be masked to the study drug. The parents of the subject, the regular staff nurses and doctors working in the unit and the project coordinator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene blue (Experimental): Subjects in the intervention arm will receive a 1 mg/kg bolus of methylene blue over 30 minutes, followed by an infusion of 0.15 mg/kg/h. The infusion rate may be increased in steps of 0.15 mg/kg/h every 30 minutes until a maximum of 0.5 mg/kg/h.
  Interventions: Drug: Methylene Blue
- Placebo infusion (Placebo Comparator): Subjects in the control arm will receive a placebo infusion (normal saline) at the same volumetric rate.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylene Blue — Subjects in the intervention arm will receive a 1 mg/kg bolus of methylene blue over 30 minutes, followed by an infusion of 0.15 mg/kg/h. The infusion rate may be increased in steps of 0.15 mg/kg/h every 30 minutes until a maximum of 0.5 mg/kg/h.
  Other Names: MB
  Arms: Methylene blue
Other: Placebo — Subjects in the placebo arm will receive normal saline in the same volumetric dose as methylene blue in the intervention arm
  Other Names: Normal saline
  Arms: Placebo infusion

SUMMARY:
Preterm infants (born at less than 37 weeks of pregnancy) sometimes develop a serious blood infection leading to low blood pressure, which does not respond to saline or to the standard medicines for increasing blood pressure, such as dopamine and epinephrine. The goal of this research study is to compare the effect of giving an injectable medicine called Methylene blue (MB) versus not giving MB to such preterm infants who are unresponsive to standard treatment. The main questions that this study aims to answer is:

1. Whether MB treatment reduces death to any cause as compared to no MB treatment.
2. Whether treatment with MB reduces the time to achieve normal blood pressure
3. Whether treatment with MB reduces the time to stoppage of all blood pressure medications, steroids and normal saline.
4. Whether treatment with MB improves heart function as measured by echocardiography at 24 and 48 hours.

DETAILED DESCRIPTION:
Preterm infants with definite or probable sepsis and fluid-refractory, catecholamine-resistant septic shock will be eligible for enrolment if they have no contraindication to receive MB. After obtaining parental consent, they will be stratified as per the first-line catecholamine used and randomly allocated to receive MB (bolus followed by infusion) or no MB for 24 hours. They will be observed for all-cause mortality (primary outcome), cause-specific mortality, time to achieve hemodynamic stability and adverse effects (secondary outcomes) over a 7-day period, all-cause mortality and cause-specific mortality hospital stay and duration of hospital stay.

The main questions it aims to answer are

1. To determine whether treatment with intravenous MB therapy reduces all-cause mortality when compared to no MB treatment, among preterm neonates with catecholamine-resistant septic shock
2. To compare the time to achieve therapeutic endpoints among preterm neonates with catecholamine-resistant septic shock treated with intravenous MB versus no MB
3. To compare time to stoppage of all inotrope/vasopressor treatment among preterm neonates with catecholamine-resistant septic shock treated with intravenous MB versus no MB
4. To compare echocardiographic parameters (at 24 hours after randomization) among preterm neonates with catecholamine-resistant septic shock treated with intravenous MB versus no MB

ELIGIBILITY:
Screening Criteria: preterm infants (<37 weeks, <28 days) clinically diagnosed to have septic shock will be screened for inclusion Inclusion criteria: Subjects must fulfill all the following

1. Definite/probable sepsis :Clinical syndrome of sepsis for which bedside neonatologist starts intravenous antibiotics AND either a positive culture of otherwise sterile body fluid OR presence of any 2 or more of the following five markers of sepsis: (a) C-reactive protein >10 mg/dL; (b) procalcitonin as per age-appropriate cut-off (c) total leukocyte count and absolute neutrophilic count beyond acceptable range (d) chest X-ray adjudged as pneumonia by two independent Neonatologists.
2. Shock: adapted from the definition given by Davis et al 2017

   1. Either SBP < age and gestation appropriate cut-off OR
   2. Presence of any 2 of the following 6 parameters i. HR >205/min ii. Central pulses either week OR bounding iii. CRT >3 sec OR flash refill (<1 sec) iv. skin mottled/cool OR flushed v. urine output <0.5 ml/kg/h in the preceding 6 hours vi. DBP < age and gestation appropriate cut-off
3. Fluid and catecholamine-resistant shock: received fluid boluses up to a maximum of 40 ml/kg followed by catecholamine infusion titrated up to the maximum dose. The catecholamine infusion could be either dopamine (maximum dose 20 µg/kg/min) or epinephrine (maximum dose 0.4 µg/kg/min) or norepinephrine (maximum dose 0.4 µg/kg/min).

Exclusion Criteria:

excluded if ≥1 criterion positive:

1. G6PD deficient or family history of G6PD deficiency
2. Potentially lethal malformation
3. Congenital heart disease
4. Severe acute kidney injury
5. Family history of allergy to methylene blue or food dyes

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-03-14 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality within 7 days after randomization | 7 days
  Mortality due to any cause over 7 days after randomization

SECONDARY OUTCOMES:
Time taken to achieve therapeutic end-points within 7 days after randomization | 7 days
  Time taken to achieve therapeutic end points of shock (which include capillary refill time less than 3 seconds, normal volume pulses, warm extremities, urine output greater than 1 ml/kg/h, normal sensorium, normal mean blood pressure, normal systolic blood pressure and normal diastolic blood pressure) up to 7 days after randomization.
Time taken to stop all inotrope/vasopressor treatment within 7 days after randomisation | 7 days
  Time taken for all inotrope and vasopressor therapy to finally stop up to a maximum of 7 days after randomisation
Echocardiographic fractional shortening at 24 hour after randomization | 24 hour
  Fractional shortening will be calculated on echocardiography by measuring the percentage change in the left ventricular diameter during systole at 24 hours after randomization.
Left ventricular end-diastolic diameter (LVEDD) by echocardiography at 24 hour after randomization | 24 hour
  Left ventricular end-diastolic diameter (LVEDD) will be measured in millimetres by echocardiography at 24 hour after randomization
Left ventricular end-systolic diameter (LVESD) by echocardiography at 24 hour after randomization | 24 hour
  Left ventricular end-systolic diameter (LVESD) will be measured in millimeters by echocardiography at 24 hour after randomization
Aortic diameter by echocardiography at 24 hour after randomization | 24 hour
  Aortic diameter will be measured in millimeters by echocardiography at 24 hour after randomization
Velocity time integral (LVI) by echocardiography at 24 hours after randomization | 24 hour
  Velocity time integral (LVI) will be measured in centimeters by echocardiography at 24 hours after randomization to calculate the cardiac output.
Echocardiographic fractional shortening at 48 hour after randomization | 48 hour
  Fractional shortening will be calculated on echocardiography by measuring the percentage change in the left ventricular diameter during systole at 48 hours after randomization.
Left ventricular end-diastolic diameter (LVEDD) on echocardiography at 48 hour after randomization | 48 hour
  Left ventricular end-diastolic diameter (LVEDD) will be measured in millimeters by echocardiography at 48 hour after randomization
Left ventricular end-systolic diameter (LVESD) by echocardiography at 48 hour after randomization | 48 hour
  Left ventricular end-systolic diameter (LVESD) will be measured in millimeters by echocardiography at 48 hour after randomization
Aortic diameter by echocardiography at 48 hour after randomization | 48 hour
  Aortic diameter will be measured in millimeters by echocardiography at 48 hour after randomization
Velocity time integral (LVI) by echocardiography at 48 hours after randomization | 48 hour
  Velocity time integral (LVI) be measured by echocardiography in centimeters at 48 hours after randomization to calculate the cardiac output.
Time taken to stop vasopressor treatment | 100 days
  Time taken to stop all vasopressors during hospital stay up to a maximum of 100 days
Mortality during hospital stay | 100 days
  Mortality during the period of hospital stay up to a maximum of 100 days
Serious adverse effects | 100 days
  Serious adverse effect with special reference to oliguria, gastrointestinal bleeds, abdominal distension, and bluish discoloration of skin and urine during hospital stay up to a maximum of 100 days
Septic shock-related mortality | 7 days
  Mortality attributed to septic shock up to 7 days post-randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Sourabh Dutta, MD, PhD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Anonymized, individual patient data pertaining to publications from the study which are in the public domain will be shared with other researchers planning to conduct a study, upon reasonable written request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available one year after the publication from the study for a period of 3 years
Access Criteria: To be decided

REFERENCES:
- [Result] Hotchkiss RS, Karl IE. The pathophysiology and treatment of sepsis. N Engl J Med. 2003 Jan 9;348(2):138-50. doi: 10.1056/NEJMra021333. No abstract available. PMID 12519925
- [Result] Stolk RF, Kox M, Pickkers P. Noradrenaline drives immunosuppression in sepsis: clinical consequences. Intensive Care Med. 2020 Jun;46(6):1246-1248. doi: 10.1007/s00134-020-06025-2. Epub 2020 Apr 8. No abstract available. PMID 32270211
- [Result] Stolk RF, van der Pasch E, Naumann F, Schouwstra J, Bressers S, van Herwaarden AE, Gerretsen J, Schambergen R, Ruth MM, van der Hoeven JG, van Leeuwen H, Pickkers P, Kox M. Norepinephrine Dysregulates the Immune Response and Compromises Host Defense during Sepsis. Am J Respir Crit Care Med. 2020 Sep 15;202(6):830-842. doi: 10.1164/rccm.202002-0339OC. PMID 32520577
- [Result] Levin RL, Degrange MA, Bruno GF, Del Mazo CD, Taborda DJ, Griotti JJ, Boullon FJ. Methylene blue reduces mortality and morbidity in vasoplegic patients after cardiac surgery. Ann Thorac Surg. 2004 Feb;77(2):496-9. doi: 10.1016/S0003-4975(03)01510-8. PMID 14759425
- [Result] Ismail R, Awad H, Allam R, Youssef O, Ibrahim M, Shehata B. Methylene blue versus vasopressin analog for refractory septic shock in the preterm neonate: A randomized controlled trial. J Neonatal Perinatal Med. 2022;15(2):265-273. doi: 10.3233/NPM-210824. PMID 34719443
- [Result] Otero Luna AV, Johnson R, Funaro M, Canarie MF, Pierce RW. Methylene Blue for Refractory Shock in Children: A Systematic Review and Survey Practice Analysis. Pediatr Crit Care Med. 2020 Jun;21(6):e378-e386. doi: 10.1097/PCC.0000000000002295. PMID 32453920
- [Result] Luis-Silva F, Menegueti MG, Sato L, Peres LM, Dos Reis Sepeda C, Petroski-Moraes BC, Donadel MD, Gallo GB, Jordani MC, Mestriner F, Becari C, Basile-Filho A, Evora PRB, Martins-Filho OA, Auxiliadora-Martins M. Effect of methylene blue on hemodynamic response in the early phase of septic shock: A case series. Medicine (Baltimore). 2023 Jan 27;102(4):e32743. doi: 10.1097/MD.0000000000032743. PMID 36705345
- [Result] Ibarra-Estrada M, Kattan E, Aguilera-Gonzalez P, Sandoval-Plascencia L, Rico-Jauregui U, Gomez-Partida CA, Ortiz-Macias IX, Lopez-Pulgarin JA, Chavez-Pena Q, Mijangos-Mendez JC, Aguirre-Avalos G, Hernandez G. Early adjunctive methylene blue in patients with septic shock: a randomized controlled trial. Crit Care. 2023 Mar 13;27(1):110. doi: 10.1186/s13054-023-04397-7. PMID 36915146
- [Result] Memis D, Karamanlioglu B, Yuksel M, Gemlik I, Pamukcu Z. The influence of methylene blue infusion on cytokine levels during severe sepsis. Anaesth Intensive Care. 2002 Dec;30(6):755-62. doi: 10.1177/0310057X0203000606. PMID 12500513
- [Result] Kirov MY, Evgenov OV, Evgenov NV, Egorina EM, Sovershaev MA, Sveinbjornsson B, Nedashkovsky EV, Bjertnaes LJ. Infusion of methylene blue in human septic shock: a pilot, randomized, controlled study. Crit Care Med. 2001 Oct;29(10):1860-7. doi: 10.1097/00003246-200110000-00002. PMID 11588440
- [Result] Zhang X, Gao Y, Pan P, Wang Y, Li W, Yu X. [Methylene blue in the treatment of vasodilatory shock: a Meta-analysis]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2017 Nov;29(11):982-987. doi: 10.3760/cma.j.issn.2095-4352.2017.11.005. Chinese. PMID 29151412
- [Result] Dumbarton TC, Minor S, Yeung CK, Green R. Prolonged methylene blue infusion in refractory septic shock: a case report. Can J Anaesth. 2011 Apr;58(4):401-5. doi: 10.1007/s12630-011-9458-x. Epub 2011 Jan 19. PMID 21246318
- [Result] Zhao CC, Zhai YJ, Hu ZJ, Huo Y, Li ZQ, Zhu GJ. Efficacy and safety of methylene blue in patients with vasodilatory shock: A systematic review and meta-analysis. Front Med (Lausanne). 2022 Sep 26;9:950596. doi: 10.3389/fmed.2022.950596. eCollection 2022. PMID 36237547
- [Result] Fleischmann-Struzek C, Goldfarb DM, Schlattmann P, Schlapbach LJ, Reinhart K, Kissoon N. The global burden of paediatric and neonatal sepsis: a systematic review. Lancet Respir Med. 2018 Mar;6(3):223-230. doi: 10.1016/S2213-2600(18)30063-8. PMID 29508706
- [Result] Bentzer P, Griesdale DE, Boyd J, MacLean K, Sirounis D, Ayas NT. Will This Hemodynamically Unstable Patient Respond to a Bolus of Intravenous Fluids? JAMA. 2016 Sep 27;316(12):1298-309. doi: 10.1001/jama.2016.12310. PMID 27673307
- [Result] Aya HD, Ster IC, Fletcher N, Grounds RM, Rhodes A, Cecconi M. Pharmacodynamic Analysis of a Fluid Challenge. Crit Care Med. 2016 May;44(5):880-91. doi: 10.1097/CCM.0000000000001517. PMID 26683506
- [Result] Nandhabalan P, Ioannou N, Meadows C, Wyncoll D. Refractory septic shock: our pragmatic approach. Crit Care. 2018 Sep 19;22(1):215. doi: 10.1186/s13054-018-2144-4. PMID 30231909
- [Result] Park BK, Shim TS, Lim CM, Lee SD, Kim WS, Kim DS, Kim WD, Koh Y. The effects of methylene blue on hemodynamic parameters and cytokine levels in refractory septic shock. Korean J Intern Med. 2005 Jun;20(2):123-8. doi: 10.3904/kjim.2005.20.2.123. PMID 16134766
- [Result] Evora PR, Roselino CH, Schiaveto PM. Methylene blue in anaphylactic shock. Ann Emerg Med. 1997 Aug;30(2):240. doi: 10.1016/s0196-0644(97)70152-5. No abstract available. PMID 9250657
- [Result] Kudawla M, Dutta S, Narang A. Validation of a clinical score for the diagnosis of late onset neonatal septicemia in babies weighing 1000-2500 g. J Trop Pediatr. 2008 Feb;54(1):66-9. doi: 10.1093/tropej/fmm065. Epub 2007 Aug 14. PMID 17698886
- [Result] Davis AL, Carcillo JA, Aneja RK, Deymann AJ, Lin JC, Nguyen TC, Okhuysen-Cawley RS, Relvas MS, Rozenfeld RA, Skippen PW, Stojadinovic BJ, Williams EA, Yeh TS, Balamuth F, Brierley J, de Caen AR, Cheifetz IM, Choong K, Conway E Jr, Cornell T, Doctor A, Dugas MA, Feldman JD, Fitzgerald JC, Flori HR, Fortenberry JD, Graciano AL, Greenwald BM, Hall MW, Han YY, Hernan LJ, Irazuzta JE, Iselin E, van der Jagt EW, Jeffries HE, Kache S, Katyal C, Kissoon N, Kon AA, Kutko MC, MacLaren G, Maul T, Mehta R, Odetola F, Parbuoni K, Paul R, Peters MJ, Ranjit S, Reuter-Rice KE, Schnitzler EJ, Scott HF, Torres A Jr, Weingarten-Abrams J, Weiss SL, Zimmerman JJ, Zuckerberg AL. The American College of Critical Care Medicine Clinical Practice Parameters for Hemodynamic Support of Pediatric and Neonatal Septic Shock: Executive Summary. Pediatr Crit Care Med. 2017 Sep;18(9):884-890. doi: 10.1097/PCC.0000000000001259. No abstract available. PMID 28723883
- [Result] Zubrow AB, Hulman S, Kushner H, Falkner B. Determinants of blood pressure in infants admitted to neonatal intensive care units: a prospective multicenter study. Philadelphia Neonatal Blood Pressure Study Group. J Perinatol. 1995 Nov-Dec;15(6):470-9. PMID 8648456
- [Result] Kermorvant-Duchemin E, Laborie S, Rabilloud M, Lapillonne A, Claris O. Outcome and prognostic factors in neonates with septic shock. Pediatr Crit Care Med. 2008 Mar;9(2):186-91. doi: 10.1097/PCC.0b013e31816689a8. PMID 18477932
- [Result] Baske K, Saini SS, Dutta S, Sundaram V. Epinephrine versus dopamine in neonatal septic shock: a double-blind randomized controlled trial. Eur J Pediatr. 2018 Sep;177(9):1335-1342. doi: 10.1007/s00431-018-3195-x. Epub 2018 Jun 23. PMID 29936590
- See also: Global report on the epidemiology and burden of sepsis [Internet]. 2020 — https://www.who.int/publications/i/item/9789240010789

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT06306001/Prot_SAP_000.pdf